CLINICAL TRIAL: NCT02280850
Title: Efficacy and Safety Study of Guanxin Shutong Capsule to Treat Chronic Stable Angina: A Randomised, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Safety Study of Guanxin Shutong Capsule to Treat Chronic Stable Angina
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaanxi Buchang Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YL-CTP-Z20020055
Record Dates: First submitted 2014-10-23; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Angina, Stable
Keywords: Angina
MeSH Terms: conditions — Angina, Stable; Angina Pectoris | interventions — guanxin shutong; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guanxin Shutong Capsule (Experimental): 3 capsules once, tid, Oral Duration: 4 weeks
  Interventions: Drug: Guanxin Shutong Capsule; Drug: nitroglycerine
- Placebo Capsule (Placebo Comparator): Placebo capsule and Guanxin Shutong Capsule the same appearance are made by SHAANXI BUCHANG PHARMACEUTICAL CO.,LTD.
  3 capsules once, tid, Oral Duration: 4 weeks
  Interventions: Drug: Placebo Capsule; Drug: nitroglycerine

INTERVENTIONS:
Drug: Guanxin Shutong Capsule — 3 capsules three times a day; Duration: 4 weeks. Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: Guanxin Shutong Capsule
Drug: Placebo Capsule — 3 capsules three times a day; Duration: 4 weeks.
  Arms: Placebo Capsule
Drug: nitroglycerine — Adults: 0.25mg-0.5mg (half pill or 1 pill) once, sub-lingual. One more pill per 5 minutes untill pain relief. If total dose is 3 pills in 15 minutes and the pain is still in, please seek medical advice urgently.
  The participators in both arms who have agina symptom will take Nitroglycerine. So the accumulated consumption of participators is the one of the maesuremnts.

SUMMARY:
Compared with placebo, assess of the efficacy and safety of Guanxin Shutong capsule to treat chronic stable angina (syndrome of blood stasis resistance), and the result will be used for the basis of later Ⅳ clinical trial.

DETAILED DESCRIPTION:
1. Procedures 1.1 Start-up stage (-14~0 Day)

1. Inquire medical history, medication use, accompanied treatment, etc;
2. Sign informed consent;
3. Measure vital signs and conduct physical examination;
4. Record symptom and signs;
5. Confirm inclusion/exclusion criteria, and put patients who meet inclusion criteria into start-up stage;
6. Record participators' history of angina pectoris and treatment, or select stable angina from outpatient service (without medicate);
7. Allocate screen number, hand out Guanxi Shutong Capsules Placebo and record card of angina/nitroglycerin used;
8. Advise patient return visit with an empty belly 2 weeks later. 1.2 Interview 1 (Baseline 0 Day)

(1) Measure vital signs; (2)Accomplish all the examination items: Blood routines, Urine routines, Stool routines + Occult blood, Hepatorenal function (AST, ALT, TBIL, ALP, γ-GT, BUN, Cr), Four coagulation tests (TT, PT, APTT, FIB), Blood fat (TC, TG, HDL-C, LDL-C), 12 leads electrocardiogram, Seattle Angina Ques-tionnaire (SAQ). Additionally, premenopausal women receive urine pregnancy test; (3) Exercise treadmill testing (ETT): around am. 10:00 (Note: Just for the patients who need ETT); (4) Record symptoms and signs ( Score of syndrome of Chinese medicine and Score of angina); (5) Randomize and allocate drug number; (6) Hand out the drugs for 2 weeks and record card of angina/nitroglycerin used; (7) Advise patient return visit 2 weeks later. 1.3 Interview 2 (14±2 Day)

1. Inquire adverse events;
2. Inquire accompanied treatment and record combined medication.
3. Measure vital signs;
4. Record symptoms and signs (Score of syndrome of Chinese medicine and Score of angina);
5. Withdraw remained drugs and box, and record card;
6. Hand out the drugs for 2 weeks and record card of angina/nitroglycerin used;
7. Advise patient return visit 2 weeks later. 1.4 Interview 3 (28±2 Day)

(1) Inquire adverse events; (2) Inquire accompanied treatment and record combined medication. (3) Measure vital signs; (4) Record symptoms and signs (Score of syndrome of Chinese medicine and Score of angina); (5) 12 leads electrocardiogram (6) Accomplish all the examination items: Blood routines, Urine routines, Stool routines + Occult blood, Hepatorenal function (AST, ALT, TBIL, ALP, γ-GT, BUN, Cr), Four coagulation tests (TT, PT, APTT, FIB), Blood fat (TC, TG, HDL-C, LDL-C), 12 leads electrocardiogram, Seattle Angina Ques-tionnaire (SAQ); (7) Exercise treadmill testing (ETT) (Note: Just for the patients who need ETT); (8) Withdraw remained drugs and box, and record card; (9) Assess compliance; (10) Summarize the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Symptom of chronic stable angina is sustained for 3 months or over 3 months (typical symptoms of myocardial ischemia occurred at least 2 times in the latest week, and angina type is stable angina (Canada CCS class Ⅰ、Ⅱ or Ⅲ);
* Blood stasis resistance on traditional Chinese medicine syndrome differentiation;
* Patients who meet the following any situation:

  1. had coronary angiography and verified a least one main branch of coronary stenosis ≥50%;
  2. have typical angina symptom, and also have positive ETT result or CTA shows at least one main branch of coronary stenosis ≥50%;
  3. had history of myocardial infarct (at least 6 months).
* Written informed consent.

Exclusion Criteria:

* Acute coronary syndrome or highly suspected acute coronary syndrome;
* Variant angina or unstable angina;
* Myocardial infarction within the past 6 months;
* Left main disease and without revascularization was verified through angiography or CTA;
* Moderate to severe aortic stenosis, hypertrophic Obstructive Cardiomyopathy or congestive heart-failure (NYHA class Ⅲ-Ⅳ);
* Patients who were received PCI/CABG within 1 year;
* Patients who are poor control of high blood pressure (SBP>170mmHg, or DBP>100mmHg);
* Patients who have hypotension (SBP<90mmHg, DBP<60mmHg) or had orthostatic hypotension;
* ECG shows complete left bundle branch block, pre-excitation syndrome, left ventricular hypertrophy or pacemaker rhythm;
* Hypohepatia (ALT or bilirubin level is higher than upper limit), renal insufficiency (serum creatinine level is higher than upper limit);
* Active peptic ulcer or skin ulcer;
* Diagnosed chest pain caused by severe neurosis, menopausal syndrome, hyperthyroidism, cervical spondylosis, gallbladder-cardiac syndrome, gastroesophageal reflux, esophageal hiatus hernia or in aortic dissection;
* Patients had hematological disorder, specific bleeding or warfarin caused bleeding;
* Drug abuser, patients with history of alcoholism in the past 2 years or dependency to known drugs;
* Psychopath;
* Patients who can't compelet exercise test (note: just for partial patients who need to complete exercise test);
* Pregnancy or lactation;
* Patients who are known or suspected hypersensitive to the study medicine or allergic constitution;
* Patients who were received big surgery within 4 weeks or participated in other clinical trials within 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effect to Angina ( Average value of angina frequency) | 6 weeks
  Record angina frequency per week. Record date is Start-up Stage 1st week, Start-up Stage 2st week, Interview Stage 1st week, Interview Stage 2st week, Interview Stage 3st week and Interview Stage 4st week (Toal of 6 times).
Exercise treadmill testing (ETT) | 4 weeks
  ST-segment displacement in electrocardiogram: Observe ST-segment displacement of J point after 60ms, including the degree of ST-segment depression.

SECONDARY OUTCOMES:
Usage of nitroglycerine per day (average value) | 4 weeks
Seattle Angina Ques-tionnaire (SAQ) | 4 weeks
Scores on Chinese medical syndrome scale | 4 weeks
  Primary symptom: Chest pains (0; Slight: 2; Moderate: 4; Severe: 6) Chest congestion (0; Slight: 2; Moderate: 4; Severe: 6) Secondary symptom: Palpitation (0; Slight: 1; Moderate: 2; Severe: 3) Shortness of breath (0; Slight: 1; Moderate: 2; Severe: 3) Insomnia (0; Slight: 1; Moderate: 2; Severe: 3)
Electrocardiogram manifestation | 4 weeks
  Compare the changes of electrocardiogram manifestation (such as ST segment, T wave) of angina before and after treatment.
Time of angina break out from exercise beginning in ETT | 4 weeks
Time of ST below 1 mm from exercise beginning in ETT | 4 weeks

OTHER OUTCOMES:
Blood fat (TC, TG, HDL-C, LDL-C) | 4 weeks
Degree and duration of angina attack. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lv Shuzheng, Principal Investigator — Beijing Anzhen Hospital; Zhang Yan, Principal Investigator — The Affiliated Hospital of Liaoning Hospital of Traditional Chinese Medicine; Chen Bojun, Principal Investigator — The Second Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine; Luo Wei, Principal Investigator — Xuzhou Central Hospital; Jiang Binghua, Principal Investigator — Shandong University of Traditional Chinese Medicine; Zhang Zhenxian, Principal Investigator — Luohe Hospital of Traditional Chinese Medicine; Xing Yanjun, Principal Investigator — First Hospital of Shijiazhuang City
Locations (1):
- The General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Li Y, Zhang L, Lv S, Wang X, Zhang J, Tian X, Zhang Y, Chen B, Liu D, Yang J, Dong P, Xu Y, Song Y, Shi J, Li L, Wang X, Han Y. Efficacy and safety of oral Guanxinshutong capsules in patients with stable angina pectoris in China: a prospective, multicenter, double-blind, placebo-controlled, randomized clinical trial. BMC Complement Altern Med. 2019 Dec 11;19(1):363. doi: 10.1186/s12906-019-2778-z. PMID 31829173